



## Consent Form for Participants Able to Give Consent

Full Title of Project: The prevalence and significance of low QRS voltages in young

healthy individuals and athletes

Centre name: Royal Brompton Hospital

Study Protocol number: IRAS 283055

NCT05799833

Version: 3.0 22/06/2023



## Imperial College London Research Governance Integrity Team

## Consent Form for Participants Able to Give Consent

Centre name: Royal Brompton Hospital

Study Protocol number: IRAS 283055

NCT05799833

Version: 3.0 22/06/2023

Full Title of Project: The prevalence and significance of low QRS voltages in

young healthy individuals and athletes

Name of Principal Investigator: Dr Sabiha Gati

Please initial box/Tick Yes or No

| 1. | I confirm that I have read and understand the participant information sheet version 1.0 dated 21.07.2022 for the prevalence and significance of low QRS voltages in young healthy individuals and athletes project and have had the opportunity to ask questions which have been answered fully. | |
|---|---|---|
| 2. | I understand that my participation is voluntary, and I am free to withdraw at any time, without giving any reason and without my legal rights nor treatment / healthcare being affected. | |
| 3. | I understand that sections of any of my medical notes may be looked at by responsible individuals from Royal Brompton Hospital, from NHS Trust or from regulatory authorities where it is relevant to my taking part in this research. | |
| 4. | I give consent for information collected about me to be used to support other research or in the development of a new test, medication, medical device or treatment (delete as applicable) by an academic institution or commercial company in the future, including those outside of the United Kingdom (which Imperial has ensured will keep this information secure). | YES □<br>NO □ |
| 5. | I give consent for samples (human tissue) collected about me<br>to be used to support other research or in the development of<br>a new test, medication, medical device or treatment (delete<br>as applicable) by an academic institution or commercial | YES □<br>NO □ |



## Imperial College London Research Governance Integrity Team

| | company in the future, inc<br>Kingdom (which Imperial h<br>information secure). | | | |
|---|---|---|---|---|
| 6. | I understand that tissue same are a gift donated to In personally benefit financia invention and/or the succemedication treatment, production | | | |
| 7. | ance of<br>d | | | |
| 8. | . I give consent to being contacted about the possibility to take part in other research studies. | | | YES □<br>NO □ |
| 9. | YES □<br>NO □ | | | |
| 10 | YES □<br>NO □ | | | |
| Name of participant | | Signature | Date | |
| Name of person taking consent (if different from Principal Investigator) | | Signature | <br>Date | |
| 1 copy for participant: 1 copy for Principal Investigator 1 copy for hospital notes | | | | |

To ensure confidence in the process and minimise risk of loss, all consent forms must be printed, presented and stored in double sided format